CLINICAL TRIAL: NCT05297968
Title: Study on the Human Bioequivalence of Oseltamivir Phosphate For Oral Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QL-ASTWOS-001
Record Dates: First submitted 2022-01-28; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Oseltamivir; Suspensions

STUDY DESIGN:
Intervention Model Description: randomized,two-treatment,two-period,two-sequence
Masking Description: open
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oseltamivir Phosphate For Oral Suspension/Tamiflu (Active Comparator): Tamiflu ,6mg/ml,batch no.3235821,manufactured by F.Hoffmann-La Roche Ltd.
  Interventions: Drug: Oseltamivir Phosphate For Oral Suspension/Tamiflu
- Oseltamivir Phosphate For Oral Suspension (Experimental): 6mg/ml,batch no.GH1A0003,manufactured by Qilu Pharmaceutical(Hainan) Co., Ltd.
  Interventions: Drug: Oseltamivir Phosphate For Oral Suspension

INTERVENTIONS:
Drug: Oseltamivir Phosphate For Oral Suspension/Tamiflu — the subjects randomly received single oral administration of Oseltamivir Phosphate For Oral Suspension/Tamiflu 75mg (6mg/ml,12.5ml)
  Other Names: tamiflu
  Arms: Oseltamivir Phosphate For Oral Suspension/Tamiflu
Drug: Oseltamivir Phosphate For Oral Suspension — the subjects randomly received single oral administration of Oseltamivir Phosphate For Oral Suspension 75mg (6mg/ml,12.5ml)
  Arms: Oseltamivir Phosphate For Oral Suspension

SUMMARY:
an open label,balanced,randomized,two-treatment,two-period,two-sequence,single dose,crossover,oral bioequivalence Study of oseltamivir phosphate for oral suspension in healthy ,adult,human subjects under fasted/fed conditions.

DETAILED DESCRIPTION:
72 healthy adult subjects will be enrolled and randomized in the study.In each period,total 21 venous blood samples (3ml each)will be collected at 0h，10min,20min,30min,45min,1h,1.25h,1.5h,1.75h,2h,2.25h,2.5h,3h,3.5h,4h,4.5h,5h,6h,8h,12h,24h,36h.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects are able to give the signed ICF before the study, and fully understand the study content, process and possible adverse reactions; 2) Subjects are able to complete the study in compliance the study in compliance with the protocol; 3) Subjects (including male subjects) agree to adopt effective contraceptive methods and not plan to get pregnant or to donate sperm or ovum from 14 days before screening to 3 months after study completion; 4) Healthy male and female subjects above 18 years of age ( inclusive); 5) Male subjects who are at least 50 kg and female subjects who are at least 45 kg, with a Body Mass Index (BMI)= Weight/Height2 (kg/m2) between 19.0-26.0 kg/m2 (both inclusive);

Exclusion Criteria:

1. History of specific allergies (asthma, etc.), allergies (such as those who are allergic to two or more drugs, foods such as milk or pollen), or hypersensitivity to Oseltamivir Phosphate or any excipients or related class of drugs
2. People with rare hereditary galactose intolerance or fructose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption or sucrase-isomaltase deficiency;
3. No history of cardiac, hepatic, renal, digestive tract, nervous system, mental and metabolic disorders, etc.;
4. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption;
5. History of surgery within 3 months prior to first dosing;
6. 5 or more cigarettes per day on average within 3 months before the screening;
7. Use of any drugs within 14 days prior to dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-27 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | up to 1 year
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-t) | up to 1 year
  Evaluation of Area under the plasma concentration versus time curve (AUC0-t)
Area under the plasma concentration versus time curve (AUC0-∞) | up to 1 year
  Evaluation of Area under the plasma concentration versus time curve (AUC0-∞)
Bioequivalence | up to 1 year
  Analysis of variance (ANOVA) was performed after logarithmic conversion of main pharmacokinetic parameters (Cmax, AUC) to calculate 90% confidence interval of geometric mean ratio of main pharmacokinetic parameters of the two preparations, and equivalence comparison was conducted. The equivalent interval was set to 80.00%~125.00%

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 1 year
  Collection of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: yu Cao, Dr, Principal Investigator — the study director of phase I clinical research center
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No